CLINICAL TRIAL: NCT03759522
Title: Assessment of Neuroinflammation in Central Inflammatory Disorders Using [F-18]DPA-714.
Acronym: DPA-714
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R18-118
Record Dates: First submitted 2018-11-06; First posted 2018-11-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome; Multiple Sclerosis; Healthy
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Controls (Experimental)
  Interventions: Drug: DPA-714 PET/MRI
- Fibromyalgia Subjects (Experimental)
  Interventions: Drug: DPA-714 PET/MRI
- Chronic Fatigue Syndrome Subjets (Experimental)
  Interventions: Drug: DPA-714 PET/MRI
- Multiple Sclerosis Subjects (Experimental)
  Interventions: Drug: DPA-714 PET/MRI

INTERVENTIONS:
Drug: DPA-714 PET/MRI — DPA-714 PET/MRI

SUMMARY:
The primary objective of this study is to measure the concentration and the regional brain distribution of activated brain microglia/macrophages using the PET radiopharmaceutical [F-18]DPA-714 in individuals with chronic pain and fatigue suspected to be associated with neuroinflammation. The PET tracer [F-18]DPA-714 binds to the 18 kDa translocator protein (TSPO, also known as the peripheral benzodiazepine receptor) in the mitochondria of activated microglia/macrophages and provides a non-invasive measure of neuroinflammation. The primary objective of this study is to determine if pain and fatigue patients have higher levels of neuroinflammation than HC individuals as measured with [F-18]DPA-714-PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age
2. Healthy volunteer OR Clinical diagnosis of Multiple Sclerosis (MS) OR Meets 2016 American College of Rheumatology (ACR) case definition criteria for fibromyalgia OR Meets 1994 Fukuda case definition criteria for Chronic Fatigue Syndrome

Exclusion Criteria:

1. Contraindication to MRI
2. Pregnancy
3. Lactation
4. Individuals who are unable to participate in the imaging portion due to severity of their medical condition
5. Chronic infectious disease (e.g. HIV, HCV)
6. Viral or bacterial illness requiring medical attention and/or antibiotics within 1 month of study participation
7. Diagnosis of cancer, including leukemia
8. Blood or blood clotting disorder
9. Except for individuals with MS, a diagnosis of autoimmune disease is exclusionary
10. Positive urine β-hCG test day of procedure or a serum -hCG test within 48 hours prior to the administration of [18F]DPA-714
11. Currently enrolled in a clinical trial utilizing experimental therapies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-03 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Neuroinflammation will be measured in healthy volunteers and compared to neuroinflammation in individuals with pain and fatigue, as measured with [F-18]DPA-714-PET/MRI. | 3 years
  Quantitative PET measures of TSPO binding in brain regions including cerebral cortex, thalami, and brainstem will be compared between healthy volunteers and symptomatic study participants with pain and/or fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Mueller C, Fang YD, Jones C, McConathy JE, Raman F, Lapi SE, Younger JW. Evidence of neuroinflammation in fibromyalgia syndrome: a [ 18 F]DPA-714 positron emission tomography study. Pain. 2023 Oct 1;164(10):2285-2295. doi: 10.1097/j.pain.0000000000002927. Epub 2023 Jun 15. PMID 37326674